CLINICAL TRIAL: NCT02867761
Title: RETHINC: REdefining THerapy In Early COPD for the Pulmonary Trials Cooperative
Acronym: RETHINC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, MeiLan Han, Professor, Department of Internal Medicine, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1U01HL128952-01 (NIH); 1U01HL128952 (NIH)
Record Dates: First submitted 2016-08-12; First posted 2016-08-16 (Estimated); Results first posted 2022-08-30 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-04

CONDITIONS: COPD (Chronic Obstructive Pulmonary Disease)
Keywords: COPD; Chronic Obstructive Pulmonary Disease; Pulmonary Function Tests; Current Smoker; Former Smoker; Chronic Obstructive Airway Disease; Respiratory Symptoms
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Smoking Cessation; Signs and Symptoms, Respiratory | interventions — indacaterol; Glycopyrrolate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Indacaterol/Glycopyrrolate (Active Comparator): indacaterol/glycopyrrolate 27.5/15.6 mcg inhaled twice daily for 12 weeks
  Interventions: Drug: Indacaterol/Glycopyrrolate
- Placebo (Placebo Comparator): Placebo 27.5/15.6 mcg inhaled twice daily for 12 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Indacaterol/Glycopyrrolate — 27.5/15.6 mcg active indacaterol/glycopyrrolate
  Arms: Indacaterol/Glycopyrrolate
Drug: Placebo — 27.5/15.6 mcg placebo
  Arms: Placebo

SUMMARY:
The study hypothesis is that symptomatic current and former smokers with spirometric values within the normal range (post-bronchodilator FEV1/FVC≥0.70 and post-BD FVC ≥ 70% predicted will still derive symptomatic benefit from long-acting bronchodilator therapy even though they are excluded from current GOLD guideline recommendations.

DETAILED DESCRIPTION:
RETHINC is a 12-week multicenter, randomized, double-blind, placebo-controlled, parallel-group study to assess the efficacy and safety of indacaterol/glycopyrrolate 27.5/15.6 mcg inhaled twice daily in symptomatic current and former smokers with respiratory symptoms despite preserved spirometry as defined by CAT ≥ 10 and post-bronchodilator FEV1/FVC ratio ≥0.70, respectively.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must be able to understand and provide informed consent
2. Age 40-80
3. ≥10 pack-year smoking history
4. Post-bronchodilator FEV1/FVC ratio ≥0.70
5. Baseline CAT≥10

Exclusion Criteria:

1. Inability or unwillingness of a participant to give written informed consent or comply with study protocol.
2. Subject is pregnant, breast-feeding, or plans to become pregnant.
3. Active pulmonary infection or prior pulmonary infection where antibiotic and/or steroid treatment was completed ≤4 weeks prior to enrollment.
4. Post-BD FVC < 70% predicted
5. A primary diagnosis of asthma established by each study investigator based on ATS/ERS criteria as previously implemented in the MACRO clinical trial.
6. Known concomitant lung disease, pulmonary tuberculosis (unless confirmed by chest x-ray to be no longer active), or clinically significant bronchiectasis.
7. History (or family history) of long QT syndrome.
8. History of paroxysmal (intermittent) atrial fibrillation will be considered an exclusion. Patients with persistent atrial fibrillation as defined by continuous atrial fibrillation for at least 6 months and controlled with a rate control strategy (i.e., selective beta blocker, calcium channel blocker, pacemaker placement, digoxin or ablation therapy) for at least 6 months may be considered for inclusion. In such patients, heart rate at enrollment must be < 100/min.
9. Patients with BMI < 15 or more than 40 kg/m2.
10. Patients with diabetes Type I or uncontrolled diabetes Type II.
11. Patients who, in the judgment of the investigator, have a clinically relevant laboratory abnormality or a clinically significant condition such as (but not limited to) significant renal disease, psychiatric disease, gastrointestinal disease, unstable ischemic heart disease, arrhythmia (excluding chronic stable atrial fibrillation), uncontrolled hypertension or any other condition which in the opinion of investigator might compromise patient safety or compliance, interfere with evaluation, or preclude completion of the study.
12. Patients with any history of lung cancer.
13. Patients with narrow-angle glaucoma, symptomatic benign prostatic hyperplasia or bladder-neck obstruction or severe renal impairment or urinary retention. Benign Prostatic Hyperplasia (BPH) patients who are stable on treatment can be considered.
14. Any other past or current medical problems or findings from physical examination or laboratory testing that are not listed above, which, in the opinion of the investigator, may pose additional risks from participation in the study, may interfere with the participant's ability to comply with study requirements or that may impact the quality or interpretation of the data obtained from the study.
15. Patients with a history of hypersensitivity to any of the study drugs or to drugs from similar chemical classification, including untoward reactions to sympathomimetic amines or inhaled medication or any component thereof.
16. Patients unable to successfully use a dry powder inhaler device or perform spirometry measurements.
17. Use of other investigational drugs at the time of enrollment or within 30 days or 5 half-lives of enrollment, whichever is longer.
18. Patients receiving any protocol-specified prohibited medications..
19. Patients receiving any protocol-specified prohibited COPD related medications (will be required to undergo a required washout period prior to enrollment).

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 780 (Actual)
Dates: Start 2017-08-29 (Actual); Primary Completion 2021-07-07 (Actual); Study Completion 2021-07-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MeiLan Han, MD, MS, Principal Investigator — University of Michigan; Prescott Woodruff, MD, MPH, Principal Investigator — University of California, San Francisco
Locations (16):
- United States (16):
  - Universityof Alabama, Birmingham, Alabama
  - University of California, Los Angeles, California
  - University of California, San Francisco, California
  - LABIOMED at Harbor-UCLA Medical Center, Torrance, California
  - University of Illinois, Chicago, Illinois
  - Northwestern University, Chicago, Illinois
  - University of Iowa, Iowa City, Iowa
  - Johns Hopkins University, Baltimore, Maryland
  - University of Michigan, Ann Arbor, Michigan
  - Minneapolis VA Medical Center, Minneapolis, Minnesota
  - Minnesota Health partners, Saint Paul, Minnesota
  - Cornell University, New York, New York
  - Duke University, Durham, North Carolina
  - Temple University, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - University of Utah, Salt Lake City, Utah

REFERENCES:
- [Derived] Han MK, Ye W, Wang D, White E, Arjomandi M, Barjaktarevic IZ, Brown SA, Buhr RG, Comellas AP, Cooper CB, Criner GJ, Dransfield MT, Drescher F, Folz RJ, Hansel NN, Kalhan R, Kaner RJ, Kanner RE, Krishnan JA, Lazarus SC, Maddipati V, Martinez FJ, Mathews A, Meldrum C, McEvoy C, Nyunoya T, Rogers L, Stringer WW, Wendt CH, Wise RA, Wisniewski SR, Sciurba FC, Woodruff PG; RETHINC Study Group. Bronchodilators in Tobacco-Exposed Persons with Symptoms and Preserved Lung Function. N Engl J Med. 2022 Sep 29;387(13):1173-1184. doi: 10.1056/NEJMoa2204752. Epub 2022 Sep 4. PMID 36066078
- See also: Pulmonary Trials Cooperative website, containing information regarding RETHINC and other studies included in the Pulmonary Trials Cooperative — http://www.pulmonarytrials.org/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 780 consented, 242 were screen fails and 3 dropped out before randomization, so 535 were randomized.
Period: Overall Study
Arm/Group | Indacaterol/Glycopyrrolate | Placebo
Started | 261 | 274
Completed | 233 | 248
Not Completed | 28 | 26
Not completed — Participant withdrawn by investigator | 0 | 1
Not completed — Lost to Follow-up | 25 | 18
Not completed — Unable to complete protocol | 3 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Indacaterol/Glycopyrrolate | Placebo | Total
Number analyzed (Participants) | 261 | 274 | 535
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.6 (9.6) | 59.1 (9.8) | 58.8 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 134 | 140 | 274
  Male | 127 | 134 | 261
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 25 | 22 | 47
  Not Hispanic or Latino | 236 | 252 | 488
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 1 | 3
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 2 | 2
  Black or African American | 92 | 99 | 191
  White | 148 | 154 | 302
  More than one race | 7 | 5 | 12
  Unknown or Not Reported | 11 | 12 | 23
Region of Enrollment [Number; unit: participants]
  United States | 261 | 274 | 535
COPD Assessment Test (CAT) Score [Mean (Standard Deviation); unit: units on a scale] — 0 - 40; 0 as low symptoms (feeling better) and 40 as high symptoms (feeling worse)
  units on a scale | 17.5 (6.7) | 17.6 (6) | 17.6 (6.4)
St. George's Respiratory Questionnaire (SGRQ) Score [Mean (Standard Deviation); unit: units on a scale] — 0 - 100 score; 0 as low symptoms (feeling better) and 100 as high symptoms (feeling worse)
  units on a scale | 37.9 (21) | 38.4 (19.3) | 38.2 (20.2)
Post bronchodilator FEV1 percent predicted [Mean (Standard Deviation); unit: percent predicted] | 93.8 (14.0) | 94.9 (12.6) | 94.2 (13.3)

OUTCOME MEASURES:

1. Primary Outcome: Proportion (Percentage) of Individuals Who Experience a 4 Unit Improvement in St. George's Respiratory Questionnaire (SGRQ) at 12 Weeks and do Not Meet Criteria for Treatment Failure During the 12 Week Treatment Period
Description: Measured by units of improvement in SGRQ scores at Baseline and 12 weeks, as well as review of treatment failure status at 4 weeks and 12 weeks of treatment (treatment failure is defined by an increase in lower respiratory symptoms necessitating treatment with active, long-acting inhaled bronchodilator, corticosteroids or antibiotics).
  A 4 unit change is the minimum clinically important difference. SGRQ has a 0 - 100 score; 0 as low symptoms (feeling better) and 100 as high symptoms (feeling worse).
Time Frame: Baseline and 12 weeks
Population: In the treatment arm, 5 subjects had primary efficacy assessment >=4 weeks after the last visit that were not included in the mITT (233 - 5 = 228). One additional subject was missing SGRQ at final visit (228 - 1 = 227). In the placebo arm, 5 subjects had primary efficacy assessment >=4 weeks after the last visit that were not included in the mITT (248 - 5 = 243). An additional person did not complete final visit but had treatment failure so are still included in mITT (243 + 1 = 244).
Measure: Count of Participants; unit: Participants
Arm/Group | Indacaterol/Glycopyrrolate | Placebo
Number analyzed (Participants) | 227 | 244
Participants | 128 | 144
Statistical Analysis 1: Comparison: Indacaterol/Glycopyrrolate vs Placebo; Test type: Superiority; p = 0.65, Generalized Estimating Equation; Odds Ratio (OR) = 0.91, 95% CI 2-sided [0.60 to 1.37]

2. Secondary Outcome: Proportion of Individuals With a 2 Unit Improvement in CAT Without Treatment Failure
Description: Proportion of individuals with a 2 unit improvement in CAT without treatment failure
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Indacaterol/Glycopyrrolate | Placebo
Number analyzed (Participants) | 227 | 244
Participants | 169 | 166

3. Secondary Outcome: Proportion of Individuals With a 1 Unit Improvement in the BDI/TDI Without Treatment Failure
Description: Proportion of individuals with a 1 unit improvement in the BDI/TDI without treatment failure
Time Frame: 12 weeks
Population: Not all participants had all measures measured.
Measure: Count of Participants; unit: Participants
Arm/Group | Indacaterol/Glycopyrrolate | Placebo
Number analyzed (Participants) | 220 | 234
Participants | 80 | 80

4. Secondary Outcome: Proportion of Individuals With Both a 4 Unit Improvement in SGRQ and a 1 Unit Improvement in BDI/TDI Without Treatment Failure
Description: Measured by units of improvement in SGRQ scores at Baseline and 12 weeks, as well as review of treatment failure status at 4 weeks and 12 weeks of treatment (treatment failure is defined by an increase in lower respiratory symptoms necessitating treatment with active, long-acting inhaled bronchodilator, corticosteroids or antibiotics).
Time Frame: 12 weeks
Population: Not all participants had all measures measured.
Measure: Count of Participants; unit: Participants
Arm/Group | Indacaterol/Glycopyrrolate | Placebo
Number analyzed (Participants) | 220 | 234
Participants | 55 | 60

5. Secondary Outcome: Mean Change in St. George's Respiratory Questionnaire (SGRQ)
Description: Value at 12 Weeks Minus Baseline. SGRQ has a 0 - 100 score; 0 as low symptoms (feeling better) and 100 as high symptoms (feeling worse).
Time Frame: Baseline, 12 weeks
Population: In the treatment arm, 5 subjects had primary efficacy assessment >=4 weeks after the last visit that were not included in the mITT (233 - 5 = 228). One additional subject was missing SGRQ at final visit (228 - 1 = 227). In the placebo arm, 5 subjects had primary efficacy assessment >=4 weeks after the last visit that were not included in the mITT (248 - 5 = 243). .
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Indacaterol/Glycopyrrolate | Placebo
Number analyzed (Participants) | 227 | 243
score on a scale | -7.7 [-9.4 to -5.9] | -8.9 [-10.6 to -7.2]
Statistical Analysis 1: Comparison: Indacaterol/Glycopyrrolate vs Placebo; Test type: Superiority; p = 0.30, Linear Mixed Effects Model

6. Secondary Outcome: Mean Change in COPD Assessment Test (CAT)
Description: Value at 12 Weeks Minus Baseline. 0 - 40; 0 as low symptoms (feeling better) and 40 as high symptoms (feeling worse).
Time Frame: Baseline, 12 weeks
Population: In the treatment arm, 5 subjects had primary efficacy assessment >=4 weeks after the last visit that were not included in the mITT (233 - 5 = 228). One additional subject was missing CAT at final visit (228 - 1 = 227). In the placebo arm, 5 subjects had primary efficacy assessment >=4 weeks after the last visit that were not included in the mITT (248 - 5 = 243).
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Indacaterol/Glycopyrrolate | Placebo
Number analyzed (Participants) | 227 | 243
score on a scale | -4.5 [-5.4 to -3.5] | -4.8 [-5.8 to -3.9]
Statistical Analysis 1: Comparison: Indacaterol/Glycopyrrolate vs Placebo; Test type: Superiority; p = 0.49, Linear Mixed Effects Model

7. Secondary Outcome: Mean Change in Baseline Dyspnea Index (BDI)/Transition Dyspnea Index (TDI)
Description: Value at 12 Weeks Minus Baseline.
Time Frame: 12 Weeks
Population: Not all participants had these measures taken.
Measure: Mean (95% Confidence Interval); unit: ratio
Arm/Group | Indacaterol/Glycopyrrolate | Placebo
Number analyzed (Participants) | 219 | 233
ratio | 0.93 [0.59 to 1.27] | 0.92 [0.59 to 1.26]
Statistical Analysis 1: Comparison: Indacaterol/Glycopyrrolate vs Placebo; Test type: Superiority; p = 0.96, Linear Mixed Effects Model

8. Secondary Outcome: Area Under the Curve (AUC) 0-3 Hours for FEV1
Description: FEV1 AUC0-3h was calculated as the area under the FEV1-time curve from 0 to 3h post-dose using the trapezoidal rule, divided by the duration (3h) to report in liters.
Time Frame: At 12 weeks, FEV1 is measured at 1-hour intervals for 3 hours
Population: Not all persons completed their lung function tests.
Measure: Mean (95% Confidence Interval); unit: liters
Arm/Group | Indacaterol/Glycopyrrolate | Placebo
Number analyzed (Participants) | 175 | 199
liters | 8.09 [7.99 to 8.20] | 7.82 [7.72 to 7.92]
Statistical Analysis 1: Comparison: Indacaterol/Glycopyrrolate vs Placebo; Test type: Superiority; p < 0.001, Linear Mixed Effects Model

9. Secondary Outcome: Change From Baseline in Trough Forced Expiratory Volume Per 1 Second (FEV1) - Absolute Value
Description: Trough FEV1 at 12 week minus trough FEV1 at baseline.
Time Frame: Baseline to 12 Weeks
Population: Not all participants had all measures measured.
Measure: Least Squares Mean (95% Confidence Interval); unit: Liters
Arm/Group | Indacaterol/Glycopyrrolate | Placebo
Number analyzed (Participants) | 198 | 205
Liters | 0.04 [0.01 to 0.08] | -0.01 [-0.04 to 0.02]

10. Secondary Outcome: Change From Baseline in 12 Hour Trough Inspiratory Capacity - Absolute Value
Description: Change from baseline in 12 hour trough inspiratory capacity - absolute value
Time Frame: Baseline
Population: Not all participants had all measures measured.
Measure: Least Squares Mean (95% Confidence Interval); unit: Liters
Arm/Group | Indacaterol/Glycopyrrolate | Placebo
Number analyzed (Participants) | 194 | 203
Liters | 0.12 [0.07 to 0.18] | 0.02 [-0.03 to 0.08]

11. Secondary Outcome: Symptoms and Rescue Medication Use Based on Daily Diary
Description: Percentage of days with symptoms (shortness of breath, chest tightness, wheezing, cough, or sputum) or use of albuterol
Time Frame: During study follow-up (Baseline to 12 weeks)
Population: Not all participants submitted complete diaries.
Measure: Mean (95% Confidence Interval); unit: percentage of days
Arm/Group | Indacaterol/Glycopyrrolate | Placebo
Number analyzed (Participants) | 198 | 210
percentage of days | 67.0 [59.0 to 75.0] | 63.6 [55.7 to 71.5]
Statistical Analysis 1: Comparison: Indacaterol/Glycopyrrolate vs Placebo; P Value for percentage of days with any symptoms (shortness of breath, chest tightness, wheezing, cough, or sputum); Test type: Superiority; p = 0.35, Linear Mixed Effects Model
Statistical Analysis 2: Comparison: Indacaterol/Glycopyrrolate vs Placebo; P Value for percentage of days with shortness of breath; Test type: Superiority; p = 0.61, Linear Mixed Effects Model
Statistical Analysis 3: Comparison: Indacaterol/Glycopyrrolate vs Placebo; P Value for percentage of days with chest tightness; Test type: Superiority; p = 0.48, Linear Mixed Effects Model
Statistical Analysis 4: Comparison: Indacaterol/Glycopyrrolate vs Placebo; P Value for percentage of days with wheezing; Test type: Superiority; p = 0.81, Linear Mixed Effects Model
Statistical Analysis 5: Comparison: Indacaterol/Glycopyrrolate vs Placebo; P Value for percentage of days with cough; Test type: Superiority; p = 0.17, Linear Mixed Effects Model
Statistical Analysis 6: Comparison: Indacaterol/Glycopyrrolate vs Placebo; P Value for percentage of days with sputum; Test type: Superiority; p = 0.64, Linear Mixed Effects Model
Statistical Analysis 7: Comparison: Indacaterol/Glycopyrrolate vs Placebo; P Value for percentage of days with use of albuterol; Test type: Superiority; p = 0.84, Linear Mixed Effects Model

12. Secondary Outcome: Treatment Failure Defined by Increase in Lower Respiratory Symptoms Necessitating Treatment With Active, Long-acting Inhaled Bronchodilator, Corticosteroids or Antibiotics
Description: Treatment failure defined by increase in lower respiratory symptoms necessitating treatment with active, long-acting inhaled bronchodilator, corticosteroids or antibiotics
Time Frame: During study follow-up (baseline to 12 Weeks)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Indacaterol/Glycopyrrolate | Placebo
Number analyzed (Participants) | 227 | 244
Participants | 5 | 9

13. Secondary Outcome: Change From Baseline in Trough FEV1 - % Predicted
Description: Trough FEV1 at 12 week minus trough FEV1 at baseline.
Time Frame: Baseline to 12 Weeks
Population: Not all participants had all measures measured.
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage of predicted number
Arm/Group | Indacaterol/Glycopyrrolate | Placebo
Number analyzed (Participants) | 198 | 205
percentage of predicted number | 2.48 [1.49 to 3.47] | -0.09 [-1.06 to 0.89]

14. Secondary Outcome: Change in FEF25-75%
Description: FEF25-75%-Forced expiratory flow over the middle one half of the FVC; the average flow from the point at which 25 percent of the FVC has been exhaled to the point at which 75 percent of the FVC has been exhaled.
Time Frame: Baseline to 12 weeks
Population: Not all participants had pulmonary function tests.
Measure: Mean (95% Confidence Interval); unit: Liters per second
Arm/Group | Indacaterol/Glycopyrrolate | Placebo
Number analyzed (Participants) | 198 | 205
Liters per second | 0.07 [0.00 to 0.15] | -0.08 [-0.15 to 0.00]

ADVERSE EVENTS:
Time Frame: During the trial, approximately 12 weeks.
Arm/Group | Indacaterol/Glycopyrrolate | Placebo
All-Cause Mortality (participants affected / at risk) | 0/261 | 0/274
Serious Adverse Events (participants affected / at risk) | 4/261 | 8/274
Other Adverse Events (participants affected / at risk) | 0/261 | 0/274
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Indacaterol/Glycopyrrolate (N=261) | Placebo (N=274)
Motor Vehicle Accident (Musculoskeletal and connective tissue disorders) | 1 | 1
Abdominal Pain (Gastrointestinal disorders) | 1 | 1
Anastomotic Ulcer (Gastrointestinal disorders) | 1 | 0
Breakthrough Seizures (Psychiatric disorders) | 1 | 0
Gastric GJ junction ulcer and posterior wall perforation (Gastrointestinal disorders) | 1 | 0
Postprocedural Intraabdominal Abscess (Gastrointestinal disorders) | 1 | 0
Chest Pain (Cardiac disorders) | 1 | 0
Sigmoid diverticulitis with small abscess (Gastrointestinal disorders) | 0 | 1
Suicide Attempt (Psychiatric disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 0
Respiratory Exacerbation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Uncontrolled hypertension (Psychiatric disorders) | 0 | 1
Acute Cholecystitis (Gastrointestinal disorders) | 1 | 0
Vitamin B12 Deficiency (Psychiatric disorders) | 0 | 1
Acute Pancreatitis (Gastrointestinal disorders) | 0 | 1
Portal Hypertension (Gastrointestinal disorders) | 0 | 1
Community Acquired Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Non-displaced Fibular Fracture (Musculoskeletal and connective tissue disorders) | 0 | 1
Kidney stone with obstruction (Renal and urinary disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-07-27): https://cdn.clinicaltrials.gov/large-docs/61/NCT02867761/Prot_SAP_000.pdf